CLINICAL TRIAL: NCT03966651
Title: A Phase I Clinical Study Evaluating the Safety of Peptide Receptor Radionuclide Therapy (PRRT) With 177Lu-DOTA0-Tyr3-Octreotate in Children With Refractory or Recurrent Neuroblastoma Expressing Somatostatin Receptors.
Brief Title: A Clinical Study Evaluating the Safety of Peptide Receptor Radionuclide Therapy (PRRT) With 177Lu-DOTA0-Tyr3-Octreotate in Children With Refractory or Recurrent Neuroblastoma Expressing Somatostatin Receptors.
Acronym: NEUROBLU 02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15 TETE 04
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Neuroblastoma
Keywords: PRRT (Peptide Receptor Radionuclide Therapy); 177Lu-DOTATATE
MeSH Terms: conditions — Neuroblastoma | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRRT with 177Lu-DOTATATE (Experimental)
  Interventions: Drug: PRRT with 177Lu-DOTATATE

INTERVENTIONS:
Drug: PRRT with 177Lu-DOTATATE — Children will receive 2 Peptide Receptor Radionuclide Therapy (PRRT) using 177Lu-DOTATATE administered intravenously at 6 weeks interval.

SUMMARY:
This study is a multicenter, open label phase I dose escalation trial designed to define the Maximum Tolerated Dose (MTD) of 177Lu-DOTATATE in children with refractory or recurrent neuroblastoma.

177Lu-DOTATATE will be delivered intravenously for 2 cycles, 6 weeks apart.

The duration of study participation of each patient will be 5 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of neuroblastoma (patients can be included whatever the results of the 123ImIBG scan).
2. Recurrent or refractory neuroblastoma following at least two prior standard treatment regimen.
3. Positive 68Ga-DOTATOC PET within 6 weeks prior to day 1 dosing. Note: PET positivity is visually defined as follow: uptake should be equivalent or higher than the liver uptake for all lesions identified by conventional neuroblastoma imaging working.
4. Patient for whom no effective conventional therapy exists.
5. a) For dose levels 1 (80 MBq/kg) & 2 (100 MBq/kg): Age > 1 year and < 18 years at the time of enrollment into the study. b) For dose level 3 (120 MBq/kg):

   - If at least one patient < 2 years old has been enrolled in one of the previous dose levels (80 or 100 MBq/kg): Age > 1 year and < 18 years at the time of enrollment into the study.

   - If no patient < 2 years old was enrolled in one of the previous dose levels (80 or 100 MBq/kg): Age ≥ 2 years and < 18 years at the time of enrollment into the study.
6. Life expectancy greater than 3 months.
7. Adequate performance Status defined as: Karnofsky or Lansky Play Performance Scale ≥ 50% (depending on patient's age).
8. Adequate recovery from major surgery prior to receiving study treatment.
9. Patients must have recovered (to CTCAE grade 1 or baseline) from any acute toxicity resulting from any prior anti-cancer treatment (except alopecia and ototoxicity).
10. Patient must have adequate organ function as defined by the following values (within 6 weeks of first dose of study treatment):

    1. Bone marrow function:

       If no bone marrow disease:

       Platelets ≥ 100 x 109/L (unsupported for 72 hours) Absolute Neutrophil Count (ANC) ≥ 0.75 x 109/L Hemoglobin > 7.5 g/dL (transfusions are allowed)

       In case of bone marrow disease:

       Platelets ≥ 75 x109/L (unsupported for 72 hours) ANC ≥0.5 x 109/L Hemoglobin > 7.5 g/dL (transfusions are allowed)
    2. Renal function:

       Serum creatinine ≤1.5 ULN for age; if higher, a calculated Glomerular Filtration Rate (GFR) (2009 Schwartz formula*) must be ≥ 60 ml/min/1.73 m2

       * eGFR (mL/min/1,73 m²) = height (cm) x 36,5 / serum creatinine (µmol/L)
    3. Liver function:

       AST and ALT ≤2.5 ULN and total bilirubin ≤1.5 ULN. In case of liver metastases, AST and ALT ≤5 ULN and total bilirubin ≤2.5 ULN
    4. Cardiac function: Shortening fraction ≥ 28% or ejection fraction ≥ 55% by echocardiogram, with no clinical congestive heart failure associated. Normal pulmonary artery pressure.
11. Patient assent and patients/parent(s)/legal guardian(s) written informed consent that is consistent with French law and ICH-GCP guidelines.
12. Patients with reproductive potential (girls post menarche and males after 1st ejaculation) and sexually active must agree to practice effective contraceptive measures for the duration of study drug therapy and for at least 7 months (for females) or 4 months (for males) after completion of study drug therapy (in accordance with CTFG guidelines).
13. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Children with negative 68Ga-DOTATOC PET.
2. Chemotherapy within 4 weeks prior to the start of study treatment, high dose chemotherapy with stem cell transplantation within 3 months prior to start study treatment, long acting somatostatin analogues within 30 days prior to start of study treatment, biological therapy or investigational agents within 4 weeks prior to the start of study treatment or prior to passing 5 half-lives, i.e. systemic clearance, whatever comes first.
3. Any previous molecular radiotherapy (PRRT, 131ImiBG or other)
4. External Beam Radiation (EBR) therapy within 30 days before starting study treatment.
5. Prior extensive EBR therapy:

   * to more than 25% of the bone marrow;
   * for two kidneys : D50% (Right+ left kidneys) ≥15Gy and D30% (Right+ left kidneys) ≥ 20Gy" ; In case of a single remaining kidney (D50% ≥ 15Gy)
6. Known brain metastases, unless these metastases have been treated and stabilized for at least 3 months prior to enrolment in the study. Patients with a history of brain metastases must have a head CT or MRI with contrast to document stable disease prior to enrolment in the study.
7. Other known co-existing malignancies.
8. Hypersensitivity to 177Lu-DOTATOC, amino acid solution or 68GaDOTATATE.
9. Pre-existing clinically significant hyperkalemia not adequately corrected.
10. Participation in another study with an experimental molecule and/or procedure within 1 month prior to the first dose of experimental treatment.
11. Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study.
12. Childbearing or lactating patient.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose (MTD) of 177Lu-DOTATATE | 6 weeks for each patient

SECONDARY OUTCOMES:
Safety will be evaluated using National Cancer Institute Common Terminology Criteria for Adverse Events | 5 months for each patient

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Pellegrin, Bordeaux
  - CHU Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Reims, Reims
  - CHU Strasbourg, Strasbourg
  - CHU de Toulouse - Hôpital des enfants, Toulouse
  - IUCT-O, Toulouse